CLINICAL TRIAL: NCT02900014
Title: Validation of a Production Method of Stem Cell Isolated From the Nasal Cavity for an Innovative Cell Therapy of Cleft Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-12; 2015-A00984-45 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children with cleft (Experimental)
  Interventions: Procedure: sampling mesenchymal stem cells

INTERVENTIONS:
Procedure: sampling mesenchymal stem cells — nasal mesenchymental stem cells are collected in patients with cleft undergoing general anesthesia, during the initial surgical management of cleft

SUMMARY:
Cell therapy appears to be an alternative to treat bone defects. Scientific advances have shown in animal models and in humans that mesenchymal stem cells were good candidates to support cellular bone regeneration after transplantation. However, their collection requires invasive sampling usually bone marrow. A new candidate stem cells able to stimulate bone regeneration has recently been identified in the nasal cavity, these cells are called "ecto-mesenchymal" cells. These stem cells have very similar biological characteristics of mesenchymal stem cells of bone marrow. They exhibit a high mitogenic activity and hold great potential for differentiation into osteoblast lineage. Given their properties and their ease of access within the nasal cavity, ecto-mesenchymal stem cells offer new prospects for cell therapy targeting bone involvement. In this context, the ecto-mesenchymal stem cells represent a nasal bone reconstruction interesting alternative in particular in indication of the cleft. They are directly and easily accessible in these children when conventional surgical reconstruction. The investigators propose in this study to validate a production method of stem cell called "ecto-mesenchymal" isolated from a biopsy of the nasal cavity of children with cleft lip and palate to be able to soon propose cell therapy innovative in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients with unilateral cleft lip and alveolar (or maxilla) or labio-maxillo-palatal, requiring surgical management of reconstruction
* Children weighing more than 2 kg

Exclusion Criteria:

* Children with concomitant pathology that might alter bone turnover: osteogenesis imperfecta, kidney failure, chronic inflammatory diseases, infections, other diseases

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
number of nasal mesenchymental stem cells | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No